CLINICAL TRIAL: NCT00355550
Title: A Double-Blind, Placebo-Controlled Study of Tricaprilin (AC-1202) Administered For Ninety Days In Subjects With Age-Associated Memory Impairment
Brief Title: Tricaprilin In Age-Associated Memory Impairment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cerecin (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KET-06-003
Record Dates: First submitted 2006-07-20; First posted 2006-07-24 (Estimated); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Age-Associated Memory Impairment
Keywords: Mild Cognitive Impairment; Cognition disorders; nutritional supplement; dietary supplement
MeSH Terms: conditions — Cognitive Dysfunction; Cognition Disorders | interventions — tricaprylin; AC-1202

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- AC-1202 (Active Comparator): Tricaprilin formulation, once daily. Administered orally
  Interventions: Drug: Tricaprilin
- Matching Placebo to AC-1202 (Placebo Comparator): Placebo formulation, once daily. Administered orally
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tricaprilin — Powder formulation will be mixed in a liquid (approximately 8 oz).
  Other Names: AC-1202
  Arms: AC-1202
Other: Placebo — Powder formulation will be mixed in a liquid (approximately 8 oz).
  Other Names: Matching placebo to AC-1202
  Arms: Matching Placebo to AC-1202

SUMMARY:
The purpose of this study is to determine whether tricaprilin, a compound that increases energy availability in the brain, improves memory in older adults with "normal" loss of memory abilities since early adult life.

DETAILED DESCRIPTION:
One physiological hallmark of aging in mammals is a decreased uptake and metabolism of glucose within the brain. The impaired glucose metabolism in the brain may contribute or exacerbate the cognitive deficits observed during normal aging. Facilitation of memory in elderly individuals occurs when glucose levels are elevated by the administration of carbohydrate. However, such a treatment poses challenges since elevated blood glucose levels are difficult to maintain and must be within a relatively narrow window, as excessive hyperglycemia is associated with cognitive impairments. The purpose of this study is to explore whether increasing levels of other substrates for the brain improves cognitive functioning in normal aged individuals with memory disorders.

Study participants will be 120 men and women aged 50-85 who have been diagnosed as having Age-Associated Memory Impairment (AAMI). During the double-blind period of the protocol, 60 participants will receive tricaprilin and 60 participants will receive a matching placebo. Tricaprilin or the matching placebo will be administered once a day for ninety days by mixing powder in 8 ounces of a liquid. Each participant will be seen six (6) times: at Screening; Baseline; treatment days Days 30, 60, 90; and 14 days after the conclusion of treatment (Day 104).

ELIGIBILITY:
Inclusion Criteria:

* Complaints that memory has declined since young adult life
* Scores on standardized tests that are at least one standard deviation below the mean score of young adults

Exclusion Criteria:

* Dementia, including Alzheimer's disease and Mild Cognitive Impairment (MCI)
* Drugs that impair cognition
* Psychiatric conditions that may impair cognition (e.g.,depression etc.)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2006-07; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Changes in Psychologix and Cogscreen Test Batteries, RAVLT (Rey Auditory Verbal Learning Test) | 90 days
Number of subjects with treatment related adverse events | 90 days
  AE incidence rate per treatment group

SECONDARY OUTCOMES:
Self-reported memory improvement | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Henderson, PhD, Study Chair — Cerecin; Thomas H. Crook III, PhD, Principal Investigator — Psychologix, Inc.; Thomas Hochadel, Pharm.D., Study Director — Advanced Research Corporation
Locations (6):
- United States (6):
  - Meridien Research, Brooksville, Florida
  - University Clinical Research-DeLand, DeLand, Florida
  - Anchor Research Center, Naples, Florida
  - Renstar Medical Research, Ocala, Florida
  - University Clinical Research Center, Pembroke Pines, Florida
  - Meridien Research, St. Petersburg, Florida

REFERENCES:
- [Background] Reger MA, Henderson ST, Hale C, Cholerton B, Baker LD, Watson GS, Hyde K, Chapman D, Craft S. Effects of beta-hydroxybutyrate on cognition in memory-impaired adults. Neurobiol Aging. 2004 Mar;25(3):311-4. doi: 10.1016/S0197-4580(03)00087-3. PMID 15123336